CLINICAL TRIAL: NCT07042126
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Ccontrolled Phase Ⅲ Clinical Trail， to Evaluate the Efficacy and Safety of 611 (Recombinant Humanized Anti-interleukin-4 Receptor Alpha IgG4 Monoclonal Antibody) in Chinese Adolescents (12 Years Old≤Age < 18 Years Old) With Moderate to Severe Atopic Dermatitis (AD)
Brief Title: Evaluation of 611 in Chinese Adolescents With Moderate to Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-611-PED-AD-III-01
Record Dates: First submitted 2025-06-06; First posted 2025-06-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — entacapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 611 (Experimental)
  Interventions: Drug: 611
- placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: 611 — Double blind treatment period : 611 600 mg/450 mg at day 1，then 300 mg subcutaneous injection Q2W thereafter until week 16 Maintenance treatment period : 611 300 mg subcutaneous injection Q2W/Q3W until week 52.（The subjects in the placebo group during the double-blind treatment period need to be given a loading dose at week 16.）
  Arms: 611
Drug: Matching placebo — Double blind treatment period : placebo subcutaneous injection Q2W until week 16.
  Arms: placebo

SUMMARY:
The primary objective of the study was to evaluate the efficacy of 611 in Chinese Adolescents with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
The maximum study duration was 64 weeks per participants, including a screening period of up to 4 weeks, a 16-week Double blind treatment period，a 36-week maintenance treatment period ，and an 8-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* The subjects and their legal guardians are able to understand and comply with the research procedures, agree to participate in the research, and sign the Informed Consent Form (ICF).
* When signing the informed consent form, the age should be ≥ 12 years old and < 18 years old, gender is not restricted, and the body weight should be ≥ 30 kg at the screening and baseline.
* During the screening process, patients were diagnosed with atopic dermatitis (AD) according to the Hanifin - Rajka criteria, and their AD medical history was evaluated by researchers to be ≥ 6 months (the diagnostic criteria are not restricted for the medical history).
* At the screening and baseline, the Eczema Area and Severity Index (EASI) score is ≥ 16 points.
* At the screening and baseline, the Investigator Global Assessment (IGA) score is ≥3 points.
* At the time of screening and baseline, the affected body surface area (BSA) by atopic dermatitis (AD) is ≥10%.
* At baseline, the weekly average score of the Numerical Rating Scale (NRS) for pruritus was ≥ 4 points.
* Subjects should have relevant medical records, other medical visit records, or other evidence within the previous year for researchers to evaluate. The subjects have poor efficacy of topical drug treatment, or are medically unsuitable for topical drug treatment.
* Be willing to use a stable dose of emollient (moisturizer) on the affected areas of atopic dermatitis (AD) twice a day for at least 7 days before randomization and continue to use it throughout the study period.
* Subjects with potential fertility (e.g., females who have experienced menarche or males who have had nocturnal emissions) must agree to avoid sexual activity or use highly effective contraceptive methods throughout the entire study period and for at least 3 months after the last dose of the medication.Subjects should have no plans for reproduction, sperm donation, or egg donation during the entire study period and for at least 3 months after the last dose of the medication.

Be able to understand and complete (either independently or with the assistance of a guardian) the research - related questionnaire filling.

Exclusion Criteria:

* Merge other skin comorbidities that may interfere with the research evaluation.
* Combined with active parasitic infections (such as helminths) or suspected parasitic infections (subjects who have excluded active infections through clinical and/or laboratory examinations before randomization can be enrolled).
* Any history of vernal keratoconjunctivitis (VKC) and atopic keratoconjunctivitis (AKC).
* Randomly select patients with any malignant tumor diagnosed within the past 5 years or currently having the disease (excluding basal cell carcinoma that has been cured for ≥ 1 year, local cutaneous squamous cell carcinoma, or carcinoma in situ of the cervix).
* The subject had a severe infection requiring intravenous antibiotics and/or hospitalization within 4 weeks before randomization, or had an active infection requiring oral antibiotics within 2 weeks before randomization, and the investigator evaluated that there might be uncontrollable risks for the subject to participate in this study.
* A history of known or suspected immunosuppression, including a history of invasive opportunistic infections (such as histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis); or those who, although the infection has resolved, are considered by the investigator to be likely to have frequent recurrences.
* Those with evidence of active tuberculosis, or those who have had active tuberculosis in the past but cannot provide sufficient evidence of treatment, or those who are judged to potentially have active tuberculosis infection based on examinations such as chest X - ray or CT, medical history, contact history, symptoms, and physical signs.
* The researchers believe that there are any diseases that are severe or unstable and may affect the safety of the subjects during the study and/or prevent the subjects from completing the study, including but not limited to cardiovascular, gastrointestinal, liver, kidney, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, and mental diseases.
* Currently receiving or having received the following treatments:

  1. Within the first 2 weeks randomly selected, patients have received topical drug treatment for atopic dermatitis (AD), such as TCS, TCI, PDE inhibitors, Janus kinase (JAK) inhibitors, etc.
  2. Within the first 4 weeks before randomization, the patients received systemic treatment with traditional Chinese medicine (TCM) of unknown nature or with therapeutic effects on AD. Or within the first 1 week before randomization, they received topical treatment with Chinese herbal medicine of unknown nature or with therapeutic effects on AD.
  3. Received systemic glucocorticoids or other immunosuppressants/immunomodulators (including but not limited to cyclosporine, mycophenolate mofetil, interferon γ [IFN-γ], JAK inhibitors, compound glycyrrhizin, azathioprine, mycophenolate mofetil, and methotrexate) randomly within the first 4 weeks or 5 half - lives (whichever is longer).
  4. Received phototherapy (including but not limited to narrow - band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen plus ultraviolet A [PUVA]), tanning beds, or any other light - emitting devices with therapeutic effects on atopic dermatitis (AD) within the first 4 weeks randomly.
  5. Randomly selected patients who had received allergen-specific immunotherapy (SIT) within the previous 6 months.
  6. Received any monoclonal antibody therapy (such as dupilumab, etc.) within the first 4 months randomly or within 5 half-lives (whichever is longer) before randomization; Received any cell - depleting agents, including but not limited to rituximab, within 6 months before randomization.
  7. As judged by the researchers, patients had no response or poor efficacy to previous treatment with anti-IL-4 and/or IL-13 drugs (such as dupilumab, etc.).
  8. Previously, 611 was used.
  9. Treatment of atopic dermatitis (AD) with prescription emollients or emollients containing additives is initiated during the screening period.
* Received live vaccines or live attenuated vaccines within the first 4 weeks before randomization.
* If any of the examination indicators before screening or randomization meet the following criteria and are judged by the researcher as unsuitable for inclusion in the study:TBIL≥1.5 ULN ;ALT/AST ≥2 ULN；Cr>1.5 ULN; blood WBC is lower than LLN, which is judged by the researcher to be clinically significant and makes the subject ineligible for the study.
* At the screening, the test results are positive for hepatitis B, positive for hepatitis C virus antibody (HCVAb), positive for human immunodeficiency virus antibody (HIVAb), and positive for serum Treponema pallidum antibody (TPAb).
* Used any investigational drugs within the first 8 weeks after randomization or 5 half-lives (whichever is longer);
* Had a history of alcohol or drug abuse within 6 months before randomization;
* Known to be allergic or intolerant to any components of the investigational drug;
* Planned or were expected to undergo major surgical operations during the study period;
* Pregnant women, women planning to become pregnant during the study period, or breastfeeding women;
* According to the investigator's judgment, the subjects were not suitable to participate in the study due to other diseases or reasons.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Eczema Area and Severity Index (EASI) - 75 Response (>= 75% Improvement in Score From Baseline) at Week 16 | Baseline, Week 16
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD
Number of Participants With Investigator's Global Assessment (IGA) Score of "0" or "1" and Improvement From Baseline of Greater Than or Equal to (>=) 2 Points From Baseline to Week 16 | Baseline to Week 16
  The IGA is an assessment instrument used to rate the severity of AD globally based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity

SECONDARY OUTCOMES:
Number of Participants With Eczema Area and Severity Index (EASI) - 75 Response (>= 75% Improvement in Score From Baseline) at each efficacy evaluation visit point except for Week 16 | Baseline, Week 60
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD
Number of Participants With Investigator's Global Assessment (IGA) Score of "0" or "1" and Improvement From Baseline of Greater Than or Equal to (>=) 2 Points From Baseline to each efficacy evaluation visit point except for Week 16 | Baseline to Week 60
  The IGA is an assessment instrument used to rate the severity of AD globally based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Number of Participants With EASI-50 (>=50% Improvement From Baseline) | Baseline to Week 60
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Number of Participants With EASI-90 (>=90% Improvement From Baseline) | Baseline, Week 60
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD
Number of Participants Who Achieved >=4 Points/ >=3 Points With Improvement From Baseline in Weekly Average of Pruritus Numerical Rating Scale (NRS) Score From Baseline | Baseline, Week 60
  Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]), higher scores indicated greater severity.

OTHER OUTCOMES:
Adverse events (AEs), measurement of vital signs，physical examination，electrocardiogram and laboratory tests at each visit | Up to 60 Weeks
  The incidence and severity of treatment emergent adverse event (TEAE), including Serious Adverse Event (SAE), as well as clinical symptoms, and any abnormalities of vital signs, physical examinations，electrocardiogram，laboratory tests and, etc.
Minimum concentration (Cmin) | Baseline to Week 60
  Minimum concentration (Cmin) of 611
Percentage of Participants With Anti-drug Antibodies and Neutralizing Antibodies | Baseline to Week 60.
  Immunogenicity assessment will be based on Anti-drug Antibodies (ADAs) response and development of Neutralizing Antibodies (NABs). Percentage is calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-drug antibodies / number of evaluable participants * 100%

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Fourth Affiliated Hospital Zhejiang University School of Medicine, Jinhua, Zhejiang
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Nanchang, Zhejiang